CLINICAL TRIAL: NCT00132548
Title: A Randomised Trial of the Efficacy and Safety of Four Drug Regimens When Used for Intermittent Preventive Treatment of Malaria in Senegalese Children
Brief Title: A Trial of Four Drug Regimens for the Prevention of Malaria in Senegalese Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institut de Recherche pour le Developpement, Senegal (Other); Cheikh Anta Diop University, Senegal (Other); Ministry of Health, Senegal (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ITCRVF02
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: Malaria; Children; Intermittent preventive treatment; Senegal
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine; Artesunate

INTERVENTIONS:
Drug: Pyrimethamine/sulfadoxine
Drug: Amodiaquine
Drug: Artesunate

SUMMARY:
A recent study has shown that the administration of a single dose of sulfadoxine/pyrimethamine plus artesunate to Senegalese children on three occasions during a short malaria transmission season reduced the incidence of clinical attacks of malaria by 86%. However, use of this drug regimen led to the selection of parasites with molecular markers of resistance to pyrimethamine and sulfadoxine. Therefore, a trial of three alternative regimens has been undertaken to see if these are as effective and safe as the drug combination used in the initial study but less likely to select for drug resistance.

DETAILED DESCRIPTION:
Background:

In countries of the Sahel and sub-Sahel, malaria transmission is highly seasonal with nearly all episodes of malaria occuring during a few months of the year. However, mortality and morbidity from malaria may be very high during this period, especially in children who are the most vulnerable group. It has been shown previously in The Gambia and elsewhere in West Africa that regular administration of anti-malarial drugs throughout the period of malaria transmission (chemoprophylaxis) reduces mortality and morbidity substantially but chemoprophylaxis is difficult to sustain. Intermittent preventive treatment (IPT) differs from chemoprophylaxis in that drugs are given at less frequent intervals and drug concentrations fall below the inhibitory level between administrations. IPT was used first to protect pregnant women from malaria and this approach has proved very effective. More recently, the IPT concept has been applied to the prevention of malaria in infants, drugs being given at the same time as infant vaccines are administered. However, in areas of seasonal malaria, such as Senegal, only a small proportion of cases of severe malaria occur during the first year of life. In such areas, older children require protection. Intermittent preventive treatment in children (IPTc) is a potential way of doing this. IPTc involves the administration of drugs to all children in the age group at risk on two or three occasions during the period of high malaria transmission. In a recent study in Senegal it was shown that the administration of a single dose of sulfadoxine/pyrimethamine (SP) plus artesunate to children aged 6 weeks to 59 months reduced the incidence of clinical attacks of malaria by 86%. However, administration of these drugs was associated with selection of parasites with molecular markers of resistance to pyrimethamine and to sulfonamides. The aim of the new study was to investigate alternative drug regimens which might be equally effective but less likely to select for drug resistance.

Objective:

The object of the study was to find the most effective drug regimen for use in intermittent preventive treatment in children in Senegal.

Study Area:

The study was conducted in Niakhar, a rural area in central Senegal where the previous trial of IPTc had been conducted. In this area, malaria transmission is very seasonal with nearly all cases occuring during a three to four month period of the year. The entomological inoculation rate in the area is 10 infectious bites per person per year.

Study Population:

All children aged 1 - 5 years residing in the study area were eligible to join the trial.

Study Procedure:

Following village meetings, the families of all eligible children were contacted and asked if they wished their child to join the study. If they wished to do so, informed consent was obtained and the child randomised to one of four treatment arms. At the beginning and at the end of the malaria transmission season, children were examined and a finger prick blood sample was obtained for determination of haemoglobin and preparation of blood films for microscopy. A drop of blood was collected on filter paper for subsequent molecular studies.

Following initial evaluation children were treated with one of four drug regimens. These were SP + 1 dose of artesunate (the regimen used in the initial trial), SP + three doses of artesunate, SP + 3 doses of amodiaquine and 3 doses of amodiaquine and artesunate. Initial drug administration was given under observation. Treatment was repeated on two further occasions at monthly intervals. The health assistants responsible for giving drugs were not blinded to the study group but they played no further part in the trial. Staff who made observations in the field, for example on the prevalence of side effects, and laboratory staff were blind to the study code.

The incidence of clinical attacks of malaria in children in each randomisation group was measured during the period of the malaria transmission. Weekly home visits were made to detect any children who were sick and children in the study who attended one of the clinics in the study area with a febrile illness were identified.

Blood films were stained with Giemsa and examined by two microscopists. DNA was extracted from filter papers obtained from parasitaemic children and examined for mutations in the dhfr and dhps genes which are associated with resistance to pyrimethamine and sulfonamides respectively.

All serious adverse events were noted and reported to the Data Safety and Monitoring Board (DSMB). Home visits were made to the first 100 children in each arm of the trial seven days after drug administration to enquire about any side effects associated with drug administration.

Trial End-Points:

The primary end-point of the trial was the prevalence of markers of drug resistance to pyrimethamine and sulfonamides at the end of the malaria transmission season. Secondary end-points were the incidence of clinical attacks of malaria and the incidence of side effects.

Sample Size:

Sample size was calculated on the basis of a comparison of the three new drug regimens with the one used in the previous trial (SP + 1 dose of artesunate). It was assumed that about 20% of children in the SP + 1 dose of artesunate group would have Plasmodium falciparum parasitaemia at the end of the malaria transmission season providing around 100% samples for molecular studies. Assuming that the prevalence of resistance mutations at the dhfr codons 108, 59 and 51 was about 90%, 500 children would be needed in each study arm to give a trial with 90% power to detect a 20% reduction in the prevalence of resistance mutations in children receiving the new drug combinations at a 5% level of significance. Allowing for a loss to follow-up of about 10% a sample size of 2,200 was selected.

Monitoring:

The trial was monitored by a clinical monitor provided by the IPTi consortium. A DSMB reviewed the study protocol, standard operating procedures and approved the analytical plan.

ELIGIBILITY:
Inclusion Criteria:

* Ages 1 - 5 years
* Residence in the study area
* Informed consent

Exclusion Criteria:

* Known allergy to study drugs
* Chronic, underlying illness

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2200
Dates: Start 2004-06; Study Completion 2004-12

PRIMARY OUTCOMES:
Prevalence of drug resistance

SECONDARY OUTCOMES:
Incidence of clinical malaria
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Cheick Sokhna, PhD, Principal Investigator — Institut de Recherche pour le Developpement, Senegal
Locations (1):
- Institut de recherche pour le developpement, Dakar, Senegal

REFERENCES:
- [Derived] Sokhna C, Cisse B, Ba el H, Milligan P, Hallett R, Sutherland C, Gaye O, Boulanger D, Simondon K, Simondon F, Targett G, Lines J, Greenwood B, Trape JF. A trial of the efficacy, safety and impact on drug resistance of four drug regimens for seasonal intermittent preventive treatment for malaria in Senegalese children. PLoS One. 2008 Jan 23;3(1):e1471. doi: 10.1371/journal.pone.0001471. PMID 18213379
- See also: web site for the IPTi consortium — http://www.ipti-malaria.org